CLINICAL TRIAL: NCT00004440
Title: Study of Ibuprofen to Preserve Lung Function in Patients With Cystic Fibrosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: FDA Office of Orphan Products Development (U.S. Federal Agency)
Collaborators: Case Western Reserve University (Other)
Allocation: Randomized | Masking: None | Purpose: Treatment
Other Study IDs: 199/13438; CWRU-FDR001185
Record Dates: First submitted 1999-10-18; First posted 1999-10-19 (Estimated); Last update posted 2015-03-25 (Estimated); Status verified 2000-04

CONDITIONS: Cystic Fibrosis
Keywords: cardiovascular and respiratory diseases; cystic fibrosis; genetic diseases and dysmorphic syndromes; rare disease
MeSH Terms: conditions — Cystic Fibrosis; Respiratory Tract Diseases; Genetic Diseases, Inborn; Rare Diseases | interventions — Ibuprofen

INTERVENTIONS:
Drug: ibuprofen

SUMMARY:
OBJECTIVES:

I. Determine the effect of different doses of ibuprofen on neutrophil (polymorphonuclear leukocyte; PMN) delivery to a mucosal surface (the oral mucosa) in patients with cystic fibrosis and healthy controls.

II. Determine the duration of effect (and possible rebound effect) of ibuprofen on PMN delivery to a mucosal surface in these patients.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE:

This is an open label study. Patients are randomized into 5 arms, each consisting of 10 healthy volunteers and 5 patients with cystic fibrosis, based on the amount of ibuprofen received during the treatment period.

The study period lasts for at least 15 days and consists of 3 periods: baseline (days 1-3), treatment (days 3-12), and recovery (days 13-15 or longer). During the treatment period patients receive ibuprofen orally every 12 hours (except for a control arm that receives no ibuprofen).

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics--

Confirmed diagnosis of cystic fibrosis (CF) based on: Sweat chloride greater than 60 mEq/L AND Typical pulmonary and/or gastrointestinal manifestation of CF OR Healthy volunteers

--Prior/Concurrent Therapy--

At least 30 days since medications with anti-neutrophil or anti-inflammatory effect (e.g., aspirin, nonsteroidal anti-inflammatory drugs [NSAIDs], corticosteroids, macrolide antibiotics)

--Patient Characteristics--

Age: Patients with cystic fibrosis (CF): 5 and over; Healthy volunteers: 18 and over

Hematopoietic: No significant history of hematologic disease

Hepatic: No significant history of hepatic disease

Renal: No significant history of renal disease

Cardiovascular: No significant history of cardiovascular disease

Pulmonary: See Disease Characteristics

Neurologic: No significant history of neurologic disease

Other: Not pregnant; No significant history of peptic ulcer disease; Patients with CF free of any acute illness within 14 days; No prior hypersensitivity to any NSAID

Min Age: 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 75
Dates: Start 1996-08; Study Completion 1999-06

CONTACTS AND LOCATIONS:
Overall Officials: Michael W Konstan, Study Chair — Case Western Reserve University